CLINICAL TRIAL: NCT03354130
Title: Intervention Study to Identify Biomarkers of Processed Meat Intake
Brief Title: Biomarkers of Processed Meat Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PP201711-15
Record Dates: First submitted 2017-11-15; First posted 2017-11-27 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Biomarkers of Processed Meat Intake in Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Volunteers consume five different diets in a randomized cross-over dietary intervention.
Masking Description: Data analyst will know the foods consumed before samples were taken
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Tofu control (Active Comparator): Volunteers will consume a vegetarian diet containing tofu during 3 days for 5 meals in total
  Interventions: Other: Processed meat dietary intervention
- Non-processed pork diet (Experimental): Volunteers will consume a diet containing non-processed pork during 3 days for 5 meals in total
  Interventions: Other: Processed meat dietary intervention
- Bacon diet (Experimental): Volunteers will consume a diet containing bacon during 3 days for 5 meals in total
  Interventions: Other: Processed meat dietary intervention
- Sausage diet (Experimental): Volunteers will consume a diet containing sausage during 3 days for 5 meals in total
  Interventions: Other: Processed meat dietary intervention
- Dry-cured sausage diet (Experimental): Volunteers will consume a diet containing dry-cured sausage during 3 days for 5 meals in total
  Interventions: Other: Processed meat dietary intervention

INTERVENTIONS:
Other: Processed meat dietary intervention — Randomized cross-over dietary intervention with 5 different diets

SUMMARY:
The intake of processed meat products has been linked to several adverse health outcomes. However, estimation of their intake proves difficult. This study aims at identifying biomarkers of intake for processed meat products in blood and urine. For this, participants of a randomized cross-over dietary intervention will consume highly controlled diets containing non-processed pork, different processed meat products or no meat. Urine and plasma will be collected and analysed to identify sets of metabolites that are specific for the intake of the processed meat products.

DETAILED DESCRIPTION:
The intake of processed meat has been linked to several adverse health outcomes such as cancer. However, little is known about the respective effects of the single products in this diverse group.

Most epidemiological studies rely on self-reported questionnaires to assess the intake of different foods. Even though this method is relatively easy to perform, it is prone to errors such as memory biases of subjects or difficulties in estimating portion size. The use of food specific biomarkers may overcome this limitation by offering an objective quantification of dietary exposure. No biomarkers for the consumption of processed meat products have been established yet.

Twelve human healthy adults will participate in a randomized cross-over dietary intervention study and will consume three different processed meat products, fresh meat or no meat, each during 3 successive days followed by a 10-day washout period. The metabolite profile in urine and plasma samples will be analysed to find metabolites that are specific for the intake of the processed meat products.

The identification of these biomarkers in blood and urine will allow a more precise estimation of intake of different processed meat products. This will enable a more robust estimation of the risk linked to the intake of processed meat products.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-30
* Healthy

Exclusion Criteria:

* Vegetarians
* Smokers

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Plasma biomarkers of meat intake | After approx. 60 h of dietary intervention
  Plasma samples will be analysed by UPLC-MS to identify metabolites specific for processed meat intake
Urinary biomarkers of meat intake | After approx. 48 h of dietary intervention
  Urine samples will be analysed by UPLC-MS to identify metabolites specific for processed meat intake

SECONDARY OUTCOMES:
Biomarkers of meat intake in spot urine | 2 hours after the first dinner of each intervention period
  Spot urine samples will be analysed by UPLC-MS to identify metabolites specific for processed meat intake
Biomarkers of meat intake in spot urine | Approx. 12 h after the first dinner of each intervention period
  Spot urine samples will be analysed by UPLC-MS to identify metabolites specific for processed meat intake

CONTACTS AND LOCATIONS:
Overall Officials: Augustin Scalbert, PhD, Principal Investigator — International Agency for Research on Cancer
Locations (1):
- International Agency for Research on Cancer, Lyon, France

REFERENCES:
- [Derived] Li C, Imamura F, Wedekind R, Stewart ID, Pietzner M, Wheeler E, Forouhi NG, Langenberg C, Scalbert A, Wareham NJ. Development and validation of a metabolite score for red meat intake: an observational cohort study and randomized controlled dietary intervention. Am J Clin Nutr. 2022 Aug 4;116(2):511-522. doi: 10.1093/ajcn/nqac094. PMID 35754192
- [Derived] Wedekind R, Kiss A, Keski-Rahkonen P, Viallon V, Rothwell JA, Cross AJ, Rostgaard-Hansen AL, Sandanger TM, Jakszyn P, Schmidt JA, Pala V, Vermeulen R, Schulze MB, Kuhn T, Johnson T, Trichopoulou A, Peppa E, La Vechia C, Masala G, Tumino R, Sacerdote C, Wittenbecher C, de Magistris MS, Dahm CC, Severi G, Mancini FR, Weiderpass E, Gunter MJ, Huybrechts I, Scalbert A. A metabolomic study of red and processed meat intake and acylcarnitine concentrations in human urine and blood. Am J Clin Nutr. 2020 Aug 1;112(2):381-388. doi: 10.1093/ajcn/nqaa140. PMID 32492168
- [Derived] Wedekind R, Keski-Rahkonen P, Robinot N, Viallon V, Ferrari P, Engel E, Boutron-Ruault MC, Mahamat-Saleh Y, Mancini FR, Kuhn T, Johnson T, Boeing H, Bergmann M, Karakatsani A, Trichopoulou A, Peppa H, Agnoli C, Santucci de Magistris M, Palli D, Sacerdote C, Tumino R, Gunter MJ, Huybrechts I, Scalbert A. Syringol metabolites as new biomarkers for smoked meat intake. Am J Clin Nutr. 2019 Dec 1;110(6):1424-1433. doi: 10.1093/ajcn/nqz222. PMID 31559413